CLINICAL TRIAL: NCT04813458
Title: A Multi-centre Survey on Tramadol Abuse in Singapore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202007-00107
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rampant prescription of opioid has in part contributed to the ongoing worldwide opioid crisis. In the United States of America, it is estimated that death from the use of opioids outnumber death from motor vehicle accident deaths by more than 40%. Consequently, many countries such as America and Canada have drawn up guidelines pertaining to safe opioid prescribing.

Tramadol is often used by pain physicians to treat chronic pain. As it is a weak opioid and unscheduled in many countries, it is often considered to have a lower addiction potential compared to strong opioids. Despite this, the literature does reveal evidence of abuse, addiction and withdrawal - although the incidence of this is unclear.

In this study, the investigators aim to determine the prevalence of tramadol misuse in a pain clinic population. The investigators also aim to determine the real-life compliance of physicians to guidelines provided by International regulatory bodies (CDC) and the modifiable risk factors associated with tramadol misuse.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending pain clinic in Singapore General Hospital, Seng Kang General Hospital and Changi General Hospital

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attends pain clinic in SGH, SKGH and CGH.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Current Opioid Misuse Measure (COMM) | Baseline
  The primary outcome is the prevalence of Current Opioid Misuse (defined as a COMM score of 9 or greater) in the patients included in the cross-sectional study (ie patients who are on tramadol)

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  PHQ-9 measures depression with scores of 5-9, 10-14,15-19 and 20 or higher representing mild, moderate , moderate to severe and severe depression. PHQ-9 scores will be performed on all patients to determine the level of depression among patients prescribed tramadol.
General Anxiety Disorder-7 (GAD-7) | Baseline
  GAD-7 measures anxiety with scores of 5, 10 and 15 representing mild, moderate and severe anxiety. GAD-7 scores will be performed on all patients to determine the level of anxiety among patients prescribed tramadol.
Opioid Risk Tool (ORT) | Baseline
  ORT measures the risk of future opioid abuse. A score of equal or less than 3 correlates with a low risk of opioid abuse. Scores of 4 to 7 indicates moderate risk and scores above 8 represents high risk.ORT scores will be performed on all patients to determine the risk of future opioid misuse among patients prescribed tramadol.

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - Changi General Hospital, Singapore
  - Seng Kang General Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided